CLINICAL TRIAL: NCT00134186
Title: Phase II Trial of Motexafin Gadolinium for Treatment of Metastatic Renal Cell Carcinoma
Brief Title: Study of Motexafin Gadolinium for the Treatment of Renal Cell (Kidney) Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCYC-0219
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2007-03

CONDITIONS: Carcinoma, Renal Cell; Urogenital Neoplasms; Urologic Neoplasms; Kidney Neoplasms
Keywords: Kidney cancer; Renal cell carcinoma; Motexafin gadolinium
MeSH Terms: conditions — Carcinoma, Renal Cell; Urogenital Neoplasms; Urologic Neoplasms; Kidney Neoplasms | interventions — motexafin gadolinium

INTERVENTIONS:
Drug: motexafin gadolinium

SUMMARY:
The purpose of this study is to find out if renal cell (kidney) cancer that has spread to other parts of the body will respond to treatment with motexafin gadolinium (MGd).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Histologically confirmed renal cell carcinoma with clinically or pathologically confirmed progression
* Ineligible for interleukin-2 (IL-2) treatment and/or have had 2 or fewer prior treatments
* Measurable disease
* Hemoglobin ≥ 9 mg/dL
* ECOG performance status of 0, 1, or 2
* Willing and able to provide written informed consent

Exclusion Criteria:

* Inadequate bone marrow, renal and liver function by laboratory criteria

  * Absolute neutrophil count < 1500/µL;
  * Platelet count < 100,000/µL;
  * AST or ALT > 2 x upper limit of normal (ULN);
  * Alkaline phosphatase > 5 x ULN;
  * Total bilirubin > 2 x ULN;
  * Creatinine > 2.0 mg/dL.
* Evidence of central nervous system metastases within past year
* Uncontrolled hypertension
* Known history of porphyria, G6PD deficiency or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43

PRIMARY OUTCOMES:
Clinical response rate (CP, PR) to MGd in patients with confirmed progressive RCC (renal cell carcinoma)

SECONDARY OUTCOMES:
Clinical benefit rate (complete response [CR], partial response [PR], stable disease [SD])
Time to progression
Progression-free survival
Overall survival and survival at 6 and 12 months
Duration of clinical response

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, D.O., Principal Investigator — Methodist Hospital Genitourinary Oncology
Locations (1):
- Methodist Hospital, Houston, Texas, United States